CLINICAL TRIAL: NCT06583980
Title: The Efficacy of a Complex Interdisciplinary Nurse-Coordinated SELf-MAnagement Intervention for People With Substantial Impact From Their Inflammatory Arthritis: Protocol for the Randomized Pragmatic INSELMA Trial
Brief Title: INSELMA - a Randomised Controlled Trial
Acronym: INSELMA-RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Danish Center for Expertise in Rheumatology (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jette Primdahl, Professor in rheumatology rehabilitation, The Danish Center for Expertise in Rheumatology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: INSELMA
Record Dates: First submitted 2024-07-12; First posted 2024-09-04 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Axial Spondyloarthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Axial Spondyloarthritis

STUDY DESIGN:
Intervention Model Description: Experimental group and control group (usual care)
Who Masked: Investigator
Masking Description: It is not possible to blind the intervention to the participants and the healthcare professionals in this trial. To ensure blinding in the analyses, all patient participants will be given a number for reference and the person performing the statistical analyses will be blinded to allocation group. A research nurse will inform the participants about group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Each participant is assigned a coordinating rheumatology nurse. Based on an initial bio-psycho-social assessment, the nurse and the participant define up to five activities using the Patient Specific Functional Scale (PSFS) and agree on goals based on shared decision-making. The coordinating nurse provides self-management support in face-to-face, telephone or online consultations depending on the participant's needs during the following six months. At each face-to-face consultation with the nurse, the PSFS activities and the goals are evaluated. Each participant can get up to 2.5 hours of support from the nurse, up to 4 hours a physiotherapist and or occupational therapist, and 1 hour from a social worker. In addition, the coordinating nurse helps identify relevant offers in the participant's municipality. The coordinating nurse can plan up to two conferences with involved professionals. A final consultation with the coordinating nurse is held after the six-month intervention.
  Interventions: Behavioral: Interdisciplinary Nurse-coordinated self-management support for people with inflammatory arthritis and substantial disease impact
- Usual care (No Intervention): Usual care consists of planned consultations every 6-12 months by a rheumatologist or a rheumatology nurse and access to support from a rheumatology nurse by telephone. The planned consultations encompass review of blood tests, joint examinations, review of completed answers to questionnaires in DANBIO, adherence and evaluation of whether pharmacological adjustment is necessary. In addition, the planned nursing consultations sporadically encompass education in relation to management of the disease, symptoms and the pharmacological treatment. At the outpatient departments at the Danish Hospital for Rheumatic Diseases, Rigshospitalet-Glostrup and Frederiksberg Hospital, patients who have specific challenges can be offered an additional nursing consultation for non-pharmacological support. At Rigshospitalet-Glostrup it is also possible to refer a patient to see a physiotherapist and/ or an occupational therapist in the outpatient department.

INTERVENTIONS:
Behavioral: Interdisciplinary Nurse-coordinated self-management support for people with inflammatory arthritis and substantial disease impact — A coordinating rheumatology nurse who follows the participant for six months, goal setting and action planning with the nurse, opportunity for needs based support from a physiotherapist, an occupational therapist and a social worker, opportunity for interdisciplinary conferences to coordinate support to achieve the agreed upon goals and a final status consultation.
  Arms: Intervention group

SUMMARY:
Background:

Patients with inflammatory arthritis (IA) experience substantial impact of their disease despite optimal pharmacological treatment. To be able to manage these challenges effectively, patients require tailored self-management support from various professionals. We thus developed a six-month nurse-coordinated interdisciplinary self-management intervention (INSELMA), in collaboration with patients, clinicians and managers. A pilot study on the INSELMA intervention in 18 participants showed promising results. It is now relevant to test the intervention and compare it to a control group in a larger study .

Objectives:

The primary objective is to compare the efficacy of the INSELMA intervention to usual care (control group), on health related quality of life measured at baseline and end of intervention (6 months after baseline).

Key secondary objectives are to compare the short and longer-term effect of INSELMA on changes in mental well-being, anxiety, depression, fatigue, pain, sleep, physical activity, global impact of the disease, work ability, self-efficacy for managing chronic disease and pain and health literacy relative to usual care from baseline to 6 and 12 months after baseline and on quality of life from baseline to 12 months after baseline.

Method:

A pragmatic randomised trial with a two-group parallel design.

All participants will be randomly allocated to the intervention or usual care only .

Both groups will receive usual care. The INSELMA intervention group will be assigned a coordinating rheumatology nurse who performs an initial biopsychosocial assessment. Based on the assessment, the nurse and the patient agree on which activities and goals to work towards for the following six months. The coordinating nurse can refer the patient to see a physiotherapist, an occupational therapist or social worker if needed and can help identify offers in the patients' municipality.

The primary endpoint will be change in quality of life from baseline to 6 month after baseline. Key secondary outcome measures are collected to compare the effect of INSELMA on changes in mental well-being, anxiety, depression, fatigue, pain, self-efficacy for managing pain, physical function, global impact of the disease, sleep problems and acceptable symptoms relative to usual care from baseline to 6 and 12 months after baseline.

DETAILED DESCRIPTION:
Approximately 30% of patients with inflammatory arthritis (IA) experience substantial disease impact despite optimal pharmacological treatment. In this trial, autoimmune chronic inflammatory arthritis (IA) includes rheumatoid arthritis (RA), psoriatic arthritis (PsA), and axial spondyloarthritis (axSpA). IA is characterised by recurrent episodes of inflammation, swelling, and tenderness of peripheral and/or axial joints. If untreated, IA can lead to joint damage, deformities, and loss of function.

Despite a consistent focus on treating inflammation, people with IA still have unmet needs. Approximately 30% do not respond sufficiently to treatment with disease modifying drugs, and thus, they do not achieve remission or a state of low disease activity. Moreover, even patients considered to be in a state of remission or low disease activity often experience substantial physical, psychological, and social impact of IA on their everyday lives. A substantial part reports morning stiffness, pain, fatigue, sleep problems, anxiety, depressed mood as well as reduced mobility, work ability and decreased quality of life.

These people need individually tailored self-management support from various disciplines to be able to manage the challenges they experience in their everyday life. This need can be met through person centred biopsychosocial rehabilitation including self-management support from an interdisciplinary team of professionals, such as rheumatologists, nurses, physiotherapists (PTs), occupational therapists (OTs), and social worker focusing on enabling independence and a meaningful life with the best possible social participation and supported by others.

So far, the evidence for the effect of interdisciplinary biopsychosocial rehabilitation and outpatient self-management interventions to people with IA and substantial impact of their arthritis is scarce. We thus developed a novel six-month Interdisciplinary Nurse-coordinated SELf-MAnagement intervention (INSELMA) for patients with IA and substantial disease impact. The aim of this trial is to test the efficacy of the 6-months INSELMA intervention compared to usual care for people with IA and substantial disease impact in a randomised controlled trial (RCT).

The development of the INSELMA intervention followed the British Medical Research Council's updated framework for developing and test of complex interventions. Relevant stakeholders were involved (patient representatives, various health professionals from hospitals and municipalities and hospital managers). Theories underpinning the intervention are self-efficacy, Acceptance and Commitment Therapy (ACT), and health literacy (HL).

A feasibility test of the INSELMA intervention on 18 participants from Rigshospitalet-Glostrup in Copenhagen and the Danish Hospital for Rheumatic Diseases in Sønderborg has been conducted. In total 17 patients completed the intervention. Eight hours support from the health professionals (HPs) led to a tendency towards increase of the participants' quality of life, mental well-being, self-efficacy, and a decrease in symptoms of anxiety, depression, fatigue, and pain. Individual interviews with participants revealed that they experienced the INSELMA intervention as a great opportunity to reduce long-held challenges they had fought alone, until now. They experienced that the intervention was adapted to their specific needs and considered the six-month empathic and goal oriented support from the coordinating nurse and from physio- and occupational therapists, to be essential. It was important with time in between consultations to work towards the goals. The participants experienced decreased disease impact and improved self-management ability. Based on these positive results, the intervention is considered feasible, meaningful and promising. It is now relevant to test these proof of concept findings in a larger trial.

Hypothesis:

The trial is based on a two-sided superiority framework where the primary null hypothesis is that there is no immediate difference between the groups (H0: µ[I] = µ[C]) on change in health related quality of life (HRQoL) (primary outcome) measured by European Quality of life 5 Dimensions, 5 levels (EQ-5D-5L) index from baseline to end of intervention (6 months after baseline).

Data collection and management:

Disease related information and Patient Reported Outcomes will be collected using REDCap. A link to the questionnaires will be sent to the participants' electronic mailbox (e-Boks). In case a participant does not use e-Boks, the questionnaires will be sent by postal mail.

Recruitment:

Participants will be recruited from the rheumatology outpatient departments at the Danish Hospital for Rheumatic Diseases in Sønderborg, Rigshospitalet-Glostrup and Frederiksberg Hospital, Copenhagen, Denmark.

Participants are recruited through the national Danish Rheumatology Database (DANBIO) and the clinical consultations based on their response to the standard questionnaires in DANBIO. If their responses fulfil the initial inclusion criteria (age, diagnosis and response to Patient Acceptable Symptom State (PASS), VAS fatigue, -pain and global health), a popup text will appear at the screen with a short information about the opportunity for support in the INSELMA trial. If the patients are interested to hear more, they can add their telephone number. A research assistant will send written participant information to the interested patients' electronic mail box or by postal mail and contact them by phone within 10 working days to offer more information about the trial. If the patient is still interested to participate and fulfills the remaining in- and exclusion criteria, consent material is sent to the patient's e-Boks or by postal mail. After written consent is obtained, baseline questionnaires are sent to the participants the same way.

Randomisation and blinding:

The participants (N=120) will be allocated to either usual care (control group, n=60) or to the INSELMA intervention (intervention group, n=60). Participants will be allocated in ratio 1:1 in permuted blocks of 2 to 6 stratified by trial site (3 levels) and diagnosis (RA, axSpA or PsA). The randomisation sequences will be generated using REDCap.

It is not possible to blind the intervention to the participants and the healthcare professionals in this trial. To ensure blinding in the analyses, all participants will be given a number for reference and the person performing the statistical analyses will be blinded to allocation group. The research nurse will inform the participants about group allocation.

Sample size:

This superiority trial is powered to show a statistically significant difference between the participants allocated to the INSELMA intervention and those allocated to usual care. Using data from our previous feasibility study (N=17), it is estimated the EQ5D-5L VAS on a 0-100 scale at baseline to have a mean of 44 points (Standard Deviation (SD) 15) in the target population.

Target Difference: Based on an estimated minimal important difference between groups of 8.0, a SD of 15 (corresponding to a Cohen's effect size of >0.50), a statistical power of at least 80%, and a two-sided statistical significance level of 0.05, 114 patients will be required for the intention-to-treat population (i.e., 57 patients in each group). Expecting some attrition and drop-outs during the trial period, 120 patients (i.e., 60 patients in each group) will be included, potentially corresponding to a statistical power of more than 83% to detect a difference between groups in the intention-to-treat population.

Adverse events and harms:

All participants will continue usual care and will be monitored throughout the intervention period to detect any unintended events. Specific attention will be towards covering any serious adverse events, and mortalities.

Statistical analyses Descriptive statistics and measures will be stratified by group and will be reported as Means or Medians, and Standard Deviations (SDs) or Interquartile ranges depending on the empirical data distribution. Categorical Variables will be reported as absolute counts and proportions (percentages) for each group. Statistical analyses will be based on the intention to treat (ITT) principle, including all randomised participants independent of adherence etc. Missing data will be handled indirectly by using mixed effect effects models for the main analyses. The primary and key secondary continuous outcomes will be analysed according to the ITT population using repeated-measures linear mixed models, including a factor for treatment group (2 levels) and time, the interaction between both, and adjustments for baseline values and stratification factors. The responder indices will be analysed using logistic regression models, including a factor for group and adjustment for stratification factors, and conservatively assuming missing data to be from non-responders. Odds ratios with 95% CIs will be estimated and converted into approximate risk ratios, and interpreted as numbers needed to treat (NNT) when appropriate. All P values and 95% confidence intervals will be two sided. A full statistical analysis plan will be developed together with the senior trial biostatistician. The essential analyses will be available and published online at Clinicaltrials.gov before enrolment of the last participant.

Ethical considerations The trial will comply with the ethical principles described in the Helsinki Declaration. All participants will receive oral and written information about the trial before participation. After time for consideration, written informed consent is obtained. The participants are informed that they can withdraw from the trial at any time without losing any right to further treatment in the outpatient department currently and in the future. In case they wish to withdraw, they will be asked if they still agree to the use of their data in the analyses. The participants' consent gives the researchers access to relevant health information in DANBIO and the electronic medical journal to be able to conduct, monitor and control the trial.

Data are stored and managed in Open Patient data Explorative Network (OPEN), which is a safe storage and analysis environment in the Region of Southern Denmark complying with the General Data Protection Regulations and the Danish data protection law.

The trial is supported by the departmental managers at the involved hospitals and the patient representatives in the user council in the Danish Center for Expertise in Rheumatology at the Danish Hospital for Rheumatic Diseases.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Diagnosed with RA, PsA, or axSpA by a rheumatologist for at least 24 months. Connected to the rheumatology department of one of the participating hospitals for at least two years
* Answer "no" to the Patient Acceptable Symptom State (PASS) (36), "Think about all the ways your arthritis has affected you during the last 48 hours. If you were to remain in the next few months as you were during the last 48 hours, would this be acceptable to you?" or
* report ≥60 on at least one Visual Analogue Scale (VAS) (0-100) for fatigue, pain, or global assessment of the impact of the disease

Exclusion Criteria:

* Planned change or a change during the past three months in treatment with disease modifying anti-rheumatic drugs (DMARDs) or glucocorticoids.
* Participation in other studies of relevance for the outcomes in INSELMA (i.e. TRACE, WORK-ON, SPINCODE, COMFI, PLATE, KRAM-offer).
* Not able to speak and understand Danish sufficiently to participate without a translator
* Unstable psychiatric illness, cognitive impairment or other physical or mental issues that impede the ability to give informed consent to participation.
* Current alcohol or drug use disorder documented in their medical journal
* Pregnant or nursing a baby
* Planned or ongoing rehabilitation at the Danish Hospital for Rheumatic Diseases or Sano, a pain or sleep clinic
* Ongoing application for early retirement or planned surgery requiring admission
* Did not participate in the INSELMA feasibility study or is a patient research partner in INSELMA

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
EQ5D-5L VAS | Baseline, 6 and 12 months after baseline
  Health related quality of life 5 dimensions, 5 levels, visual analogue scale (0-100)

SECONDARY OUTCOMES:
WHO-5 | Baseline, 6 and 12 months after baseline
  World Health Organizations 5 mental health index (0-100, lover scores reflect lower mental well-being)
HADS | Baseline, 6 and 12 months after baseline
  Hospital Anxiety and Depression Scale (0-21, higher scores reflect higher risk for developing anxiety and depression)
BRAF-NRSv2 | Baseline, 6 and 12 months after baseline
  Bristol Rheumatoid Arthritis Fatigue Numerical Rating Scales version 2 for fatigue severity, impact and coping (0-100, higher scores reflect higher severity, impact and worse coping)
VAS pain | Baseline, 6 and 12 months after baseline
  Visual Analogue Scale Pain (0-100, higher scores reflect worse pain)
Pain self-efficacy | Baseline, 6 and 12 months after baseline
  Self-efficacy for managing pain (0-60, higher scores reflect higher degree of self-efficacy in managing pain)
MD-HAQ | Baseline, 6 and 12 months after baseline (in patients with rheumatoid arthritis and psoriatic arthritis only)
  Multi-dimensional Health Assessment Questionnaire, (0-3, higher scores reflect higher degree of physical limitations)
BASFI | Baseline, 6 and 12 months after baseline (in patients with psoriatic arthritis and axial spondyloarthritis only)
  Bath Ankylosing Spondylitis Functional Index (0-10, higher scores reflect higher degree of physical limitations)
VAS-global | Baseline, 6 and 12 months after baseline
  Patients assessment of impact of the disease Visual Analogue Scale (0-100, higher scores reflect higher impact)
ISI | Baseline, 6 and 12 months after baseline
  Insomnia Severity Index (0-28, higher scores reflect worse sleep problems)
PASS | Baseline, 6 and 12 months after baseline
  Patient Acceptable Symptom State (yes/no)
EQ5D-5L Index | Baseline, 6 and 12 months after baseline
  Health-related quality of life index for cost-effectiveness analyses

OTHER OUTCOMES:
HLQ subscales 3 and 6 | Baseline, 6 and 12 months after baseline
  Health Literacy Questionnaire subscale 3 (Actively managing my health, 5-20, higher scores reflect higher Health Literacy) and suscale 6 (Ability to actively engage with healthcare providers (5-25, higher scores reflect higher Health Literacy)
Smoking habits | Baseline, 6 and 12 months after baseline
  Present, occational, previous or never smoker, amount per day
Alcohol habits | Baseline, 6 and 12 months after baseline
  How many units do you drink per week?, How often do you drink? and How often do you drink five units or more on the same occation?

CONTACTS AND LOCATIONS:
Overall Officials: Jette Primdahl, PhD, Principal Investigator — University of Southern Denmark
Locations (3):
- Denmark (3):
  - Frederiksberg Hospital, Frederiksberg
  - Rigshospitalet-Glostrup, Glostrup Municipality
  - Danish Hospital for Rheumatic Diseases, Sønderborg

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-08-14): https://cdn.clinicaltrials.gov/large-docs/80/NCT06583980/SAP_000.pdf